CLINICAL TRIAL: NCT02328001
Title: Cost-Minimization Analysis and Its Impact on Resource Utilization After a Targeted Intervention for EGD and Colonoscopy
Brief Title: Cost-Minimization Analysis After a Targeted Intervention for EGD and Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sindhu R Kaitha, MD (Other)
Responsible Party: Sponsor-Investigator, Sindhu R Kaitha, MD, MD, University of Oklahoma
Organization: University of Oklahoma (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 4667
Record Dates: First submitted 2014-12-16; First posted 2014-12-31 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Primary Focus of the Study is Cost-minimization Analysis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intervention phase/phase 1 (No Intervention): No intervention will be applied in phase 1
- Post-intervention phase/phase 2 (Other): Intervention will be applied in phase 2 i.e; Debriefing endoscopists of the procedure accessory costs and pathology specimen costs
  Interventions: Behavioral: Debriefing endoscopists of the procedure accessory costs

INTERVENTIONS:
Behavioral: Debriefing endoscopists of the procedure accessory costs — Informing endoscopists of the number of accessories used and the dollar value of the accessories
  Arms: Post-intervention phase/phase 2

SUMMARY:
This study performs a single intervention of informing endoscopists how much the disposable accessories cost following each procedure. Following this single and simple intervention, prospective analysis of EGD and colonoscopy accessory use and pathology specimen costs will be compared to the same resource costs during a control period where endoscopists are blinded to their observation.

DETAILED DESCRIPTION:
This study is a prospective cost-identification and cost-minimization analysis of accessories used during the EGD and colonoscopy procedures. The endoscopists will be the participants under study and not the patients. The study will be conducted in two phases - pre and post-intervention phases. Each phase will include a minimum of 337 combined EGD and colonoscopy procedures and a total of upto a minimum 674 and a maximum of 1200 procedures for both phases. All consecutive patients undergoing EGD and colonoscopy will be included. For the first phase of the study, the endoscopist will not be made aware of the study and also will not be briefed at the end of the procedure with the number of accessories used during the procedure and the dollar value of the accessories. For the second phase of the study, endoscopist will be briefed by the endoscopy nursing staff after completion of each procedure about the total number of accessories used and the dollar value of the accessories used during the procedure. Once the study is completed, endoscopists will be debriefed about the study and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age of 18 or greater
* All races
* Indication for therapeutic EGD or colonoscopy
* Outpatient procedures done at OU Physicians Building endoscopy unit
* Procedure is performed by one of the observed endoscopists

Exclusion Criteria:

* Pediatric population
* Diagnostic EGD and colonoscopy procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total cost of accessory use and pathology specimen costs | Up to 5 months
  The cost of accessory and pathology specimens would be assessed immediately post-procedure during phase 2

CONTACTS AND LOCATIONS:
Overall Officials: William Tierney, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma University Physicians Building, OUPB, Endoscopy Unit, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Hogan RB, Santa-Cruz R, Weeks ES Jr, Alexander L, Hogan RB 3rd. Cost-minimization analysis of jumbo reusable forceps versus disposable forceps in a high-volume ambulatory endoscopy center. Gastrointest Endosc. 2009 Feb;69(2):284-8. doi: 10.1016/j.gie.2008.04.062. Epub 2008 Aug 23. PMID 18725156
- [Background] ASGE Technology Committee; Siddiqui UD, Banerjee S, Barth B, Chauhan SS, Gottlieb KT, Konda V, Maple JT, Murad FM, Pfau PR, Pleskow DK, Tokar JL, Wang A, Rodriguez SA. Tools for endoscopic stricture dilation. Gastrointest Endosc. 2013 Sep;78(3):391-404. doi: 10.1016/j.gie.2013.04.170. No abstract available. PMID 23948186
- [Background] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189
- [Background] Paspatis GA, Tribonias G, Konstantinidis K, Theodoropoulou A, Vardas E, Voudoukis E, Manolaraki MM, Chainaki I, Chlouverakis G. A prospective randomized comparison of cold vs hot snare polypectomy in the occurrence of postpolypectomy bleeding in small colonic polyps. Colorectal Dis. 2011 Oct;13(10):e345-8. doi: 10.1111/j.1463-1318.2011.02696.x. PMID 21689363
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514
- [Background] Leighton JA, Shen B, Baron TH, Adler DG, Davila R, Egan JV, Faigel DO, Gan SI, Hirota WK, Lichtenstein D, Qureshi WA, Rajan E, Zuckerman MJ, VanGuilder T, Fanelli RD; Standards of Practice Committee, American Society for Gastrointestinal Endoscopy. ASGE guideline: endoscopy in the diagnosis and treatment of inflammatory bowel disease. Gastrointest Endosc. 2006 Apr;63(4):558-65. doi: 10.1016/j.gie.2006.02.005. No abstract available. PMID 16564852